CLINICAL TRIAL: NCT00298454
Title: Forced Diuresis Vs Observation in Resolving Renal Failure After Haemofiltration in Critically Ill Patients (Fodorefh)
Brief Title: Forced Diuresis Versus Observation in Resolving Renal Failure After Haemofiltration in Critically Ill Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Number included has been reached
Sponsor: Frisius Medisch Centrum (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200601
Record Dates: First submitted 2006-03-01; First posted 2006-03-02 (Estimated); Last update posted 2007-04-19 (Estimated); Status verified 2007-04

CONDITIONS: Renal Failure; Critically Ill
Keywords: renal failure; oliguric; critically ill; furosemide
MeSH Terms: conditions — Renal Insufficiency; Critical Illness | interventions — Furosemide

INTERVENTIONS:
Drug: Furosemide

SUMMARY:
Intensive care patients with multiple organ dysfunction syndrome often show renal failure with the need for hemofiltration. Resolving renal failure after cessation of hemofiltration may or may not be accompanied by oliguria. Whether or not the administration of diuretics at that moment is appropriate is not known. The study randomises between furosemide or placebo when hemofiltration is stopped. Study endpoint is recovery of renal function.

DETAILED DESCRIPTION:
Introduction:

Virtually all intensive care (IC) patients with prolonged IC stay have multiple organ dysfunction syndrome. Frequently renal failure is present. The resolution of renal failure is often relatively late. After cessation of hemofiltration, oliguria may be present, at least for some time. Increasing diuresis by diuretics will probably increase clearance. As a result, intensive care stay and outcome may improve. However, diuretics might also be harmful as it is when applied in developing renal failure.

Aim of the study:

To study whether the stimulation of diuresis by furosemide when hemofiltration is stopped enhances renal recovery and secondary shortens the length of IC-stay.

Setting:

IC-patients treated at the Medical Centre Leeuwarden with MODS and renal failure are included when hemofiltration is stopped. The ICU is mixed medical and surgical, 16 beds with full time intensivists responsible for hemofiltration.

Study design:

Prospective randomised placebo controlled single centre trial.

Methods:

Inclusion criteria. Patients with mechanical ventilation in whom hemofiltration is stopped. Written informed consent must be obtained.

Excluded are patients with pre-existent serum creatinin of 150 umol/l or clearance less than 30 ml/min. Patients admitted with renal failure as the primary admission diagnosis in case acute renal failure is due to glomerulonephritis.

Creatinin clearance is measured in a 4 hour period directly after cessation of hemofiltration. The patient is then randomised for furosemide or sodium chloride. Furosemide is administered at 0.5 mg/kg/hour. Dehydration is prevented by infusing the patient the volume of their diuresis.

Daily creatinin clearance is calculated.

Primary endpoints:

1. Recovery of renal function (clearance more than 30 ml/min)
2. Stable or declining serum creatinin in case of persistent clearance less than 30 ml/min
3. Need for re-start of renal replacement therapy (metabolic acidosis, hyperkalaemia, fluid overload, uremia or uremic complications)

Secondary endpoints:

Length of stay ICU, mortality.

Poweranalysis:

36 patients per group for alpha 0.05 and beta 0.8 and 30% faster recovery of renal failure for the intervention group.

Statistical analysis:

Student t for normally distributed variables, otherwise non-parametric tests. Kaplan Meier and Cox regression for time to recovery of renal function.

ELIGIBILITY:
Inclusion Criteria:

* cessation of hemofiltration
* mechanical ventilation
* written informed consent

Exclusion Criteria:

* pre-existent renal failure
* glomerulonephritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72
Dates: Start 2005-12; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Creatinin clearance

SECONDARY OUTCOMES:
length of stay in the intensive care and hospital
intensive care and hospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: Peter van der Voort, MD, PhD, MSc, Principal Investigator — Dept of intensive care, Medical Centre Leeuwarden, PO Box 888,8901BR Leeuwarden, The Netherlands
Locations (1):
- Dept of intensive care, Medical Centre Leeuwarden, Leeuwarden, Provincie Friesland, Netherlands

REFERENCES:
- [Derived] Hashimoto H, Yamada H, Murata M, Watanabe N. Diuretics for preventing and treating acute kidney injury. Cochrane Database Syst Rev. 2025 Jan 29;1(1):CD014937. doi: 10.1002/14651858.CD014937.pub2. PMID 39878152
- [Derived] van der Voort PH, Boerma EC, Koopmans M, Zandberg M, de Ruiter J, Gerritsen RT, Egbers PH, Kingma WP, Kuiper MA. Furosemide does not improve renal recovery after hemofiltration for acute renal failure in critically ill patients: a double blind randomized controlled trial. Crit Care Med. 2009 Feb;37(2):533-8. doi: 10.1097/CCM.0b013e318195424d. PMID 19114909